CLINICAL TRIAL: NCT06310096
Title: Role of Thoracolumbar Fascia Stretching on Pain Parameters With Non-Specific Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atılım University (Other)
Collaborators: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, NAİME ULUG, Director, Atılım University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E-59394181-604.01-79277
Record Dates: First submitted 2024-02-06; First posted 2024-03-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Pain; Low Back Pain
Keywords: thoracolumbar fascia; stretching; pain threshold; temporal summation; low back pain.
MeSH Terms: conditions — Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLF fascial stretching exercise (Active Comparator): The study group received a 4-week TLF fascial stretching exercise (10 times per day) in addition to the conventional physiotherapy program, while the control group only received a conventional physiotherapy program
  Interventions: Other: TLF fascial stretching exercise
- conventional physiotherapy program (Active Comparator): The study group received a 4-week TLF fascial stretching exercise (10 times per day) in addition to the conventional physiotherapy program, while the control group only received a conventional physiotherapy program.
  Interventions: Other: conventional physiotherapy program.

INTERVENTIONS:
Other: TLF fascial stretching exercise — Relaxed lumbo-pelvic upright sitting with arms in neutral anatomical position (O'Sullivan et al., 2006). The subjects had to bend both knee flexed 90. The feet of the Participant lied flat on the ground. Trunk was in aligned position and the angle between upper body and lower body was 90. Seated position led to caudal tensioning of the pTLF via stretching of the gluteus maximus (GM)
  Seated position with passive arms elevation Seated position with passive caudal stretching of TLF through thigh elevation. The subjects had to bend both hips while keeping their feet onto a stool (30 cm high) so to pull the GM and the TLF
  Arms: TLF fascial stretching exercise
Other: conventional physiotherapy program. — hotpack, ultrasound ,Tens
  Arms: conventional physiotherapy program

SUMMARY:
Role of Thoracolumbar Fascia Stretching on Pain Parameters with Non-Specific Chronic Low Back Pain

DETAILED DESCRIPTION:
These findings demonstrate the significant impact of chronic pain on connective tissue health and highlight the importance of addressing this issue in the management of CLBP.

Chronic pain contributes to the persistence of chronic local connective tissue inflammation, resulting in fibrosis, connective tissue adhesions, and decreased mobility of the thoracolumbar fascia (TLF) in patients with chronic low back pain (CLBP).

Furthermore, an increase in TLF thickness, possibly due to structural changes in the connective tissue, is associated with pain severity.

Stretching the fascia is a crucial aspect of manual and movement therapies. The results of this study provide evidence for the effectiveness of TLF stretching in reducing pain and improving pain sensitivity in CLBP patients.

The language used was clear, objective, and value-neutral, avoiding biased, emotional, figurative, or ornamental language.

This study aimed to investigate the effect of TLF stretching on pain characteristics, including pain intensity, pressure pain threshold (PPT), temporal summation, pain sensitivity, and the impact of pain on activity in CLBP patients.

The study design was a randomized controlled trial and cross-sectional study.

Passive tone and impersonal construction were employed, and first-person perspectives were avoided unless necessary. High-level, standard language with consistent technical terms was used, and common sentence structure was adhered to.

The study was conducted from November 2023 to January 2024 and involved 30 participants with nonspecific chronic low back pain, aged 20-60 years, who were randomly assigned to either the study group (n=15; 7 men, 8 women) or the control group (n=15; 7 men, 8 women).

The study group received a 4-week TLF fascial stretching exercise (10 times per day) in addition to the conventional physiotherapy program, while the control group only received the conventional physiotherapy program. The study measured pain intensity using a 10-point numerical rating scale (NRS), pressure pain threshold (PPT), and temporal summation by an algometer (from TLF levels of lumbar 1 and 3 vertebrae (L1, L3) and 12th costa) as primary outcomes. Secondary outcomes comprised pain sensitivity assessed by the Pain Sensitivity Scale (PSS) and the effects of pain on activity measured by the Brief Pain Inventory (BPI).

ELIGIBILITY:
Inclusion Criteria:

* Those who are between the ages of 20-60 and agree to participate in the research,
* Those who have lower back pain for at least 3 months,
* Individuals who have no perception problems and can cooperate well,
* Individuals who attend regular checks and evaluations of the physiotherapy program.

Exclusion Criteria:

* -Those who have had spinal surgery,
* Those who complain of low back pain due to inflammatory, tumoral, metabolic reasons,
* Orthopedic obstacles to treatment (pes planus, genu varum, genu valgum, scoliosis, etc.) or Those with neurological problems (Multiple Sclerosis, Stroke, etc.),
* Those who have had spine or lower extremity surgery,
* Those who have another musculoskeletal disorder affecting the lower extremity,
* They are pregnant.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-11 (Estimated)

PRIMARY OUTCOMES:
Pain threshold | 12 weeks
  Pain threshold levels were analysed with algometer.
Temporal summation | 12 weeks
  With a cotton-tipped applicator, the points T12, L1 and L3 were tapped with a frequency of 1 cm/second. This is usually the site of cutaneous allodynia and trigger points. Three strokes were given at a predetermined interval. After each tap, patients were asked to rate the level of pain caused by the cotton-tipped applicator on a scale from 1 to 10.
  The primary outcome was pain level, which was scored from 1 to 10. Patients gave their responses verbally and these responses were recorded by the researcher.
NRS(Numerical rating scales) | 12 weeks
  We used a 10-point numerical rating scale (NRS) to assess the patient's current pain.

SECONDARY OUTCOMES:
Pain Sensitivity Scale (PSS) | 12 weeks
  In the questionnaire consisting of 17 questions, the patient's sensitivity to pain is measured with the pain sensitivity questionnaire. In the questionnaire with a 10-point Likert scale, the patient rates the pain experienced according to the questions asked.
Brief Pain Inventory (BPI) | 12 weeks
  The Brief Pain Inventory (BPI) scale is used to measure the effects of pain on activity, mood, walking, human relationships, sleep and enjoyment of life. It is graded on a 10-point Likert scale, with an increase in the total score indicating the negative effect of pain on the parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Naime Uluğ, PhD., Principal Investigator — ATILIM UNİVERSİTY
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)